CLINICAL TRIAL: NCT06127732
Title: Effects of Phytosterol Supplementation on Lipoprotein Subfractions and LDL Particle Quality: Primary Prevention Study
Brief Title: Phytosterol Supplementation and Lipoprotein Subfractions
Acronym: Phyto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria Cristina de Oliveira Izar, Assistant Professor of Medicine, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 042778/2017
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Hypercholesterolemia; Primary Prevention
Keywords: Phytosterols; Lipoproteins; LDL-subfractions; HDL-subfractions
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, crossover intervention study conducted with participants selected by the investigators, and invited to participate in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phytosterol (Experimental): Participants received diet plus phytosterols (2.6 g of phytosterols per day) prescribed and supplied in 650 mg gelatin capsules, to be used four capsules a day along with meals(Fitocor®, Farmoquímica, Brazil) and divided into two meals.for 12 weeks.
  Interventions: Dietary Supplement: Phytosterol supplements
- Control: diet alone (No Intervention): Participants received diet alone recommended for 12 weeks.

INTERVENTIONS:
Dietary Supplement: Phytosterol supplements — Participants were randomized into two groups to receive diet plus phytosterols (DP) for 12 weeks, followed by a 7-day washout period with a second period of intervention, where treatments were switched, and participants received diet alone (D) and were followed for another 12 weeks.
  Arms: Phytosterol

SUMMARY:
The goal of this clinical trial was to evaluate the effects of phytosterol supplementation to the diet on lipids, LDL and HDL subfractions, and on the quality of LDL in apparently healthy subjects.

The main questions it aims to answer are:

* do phytosterols reduce LDL-cholesterol and modify LDL and HDL subfractions?
* do phytosterols modify the quality of LDL?

Participants were aleatory selected to diet alone (D) or diet plus phytosterols (DP, 2.6 g divided in two doses, with meals) for 12 weeks, followed by a 7-day washout period, where treatments were switched for another 12-weeks.

DETAILED DESCRIPTION:
Military police from the ROTA (Rondas Ostensivas Tobias de Aguiar, N=60), with hypercholesterolemia in primary prevention were recruited. Of those, 27 did not meet entry criteria, 10 were excluded for not following the protocol. Twenty-three individuals were aleatory selected to diet alone (D) or diet plus phytosterols (DP, 2.6 g divided in two doses, with meals) for 12 weeks (w), followed by a 7-day washout period, where treatments were switched for another 12-w.

Study was prospective, randomized, open label, cross-over, with parallel arms and blinded endpoints.

Anthropometry, food consumption and laboratory parameters were evaluated every 12-w.

HDL and LDL subfractions were analyzed by the electrophoresis system in polyacrylamide gel (Lipoprint System®).

Plasma LDL was separated by ultracentrifugation and the quality of the LDL analyzed by nonlinear optical response (Z-scan and UV-vis spectroscopy techniques).

ELIGIBILITY:
Inclusion Criteria:

* participants of both sexes, aged >18 and <65 years, literate, in primary prevention of cardiovascular disease, with LDL-c ≥130mg/dL and <190 mg/dL and triglycerides <400 mg/dL.

Exclusion Criteria:

* secondary causes of dyslipidemia, renal (creatinine > 2mg/dL), hepatic (AST or ALT > 1.5 ULN), or metabolic (HbA1c >8.0%) dysfunction, with BMI <18.5 or >40 Kg/m2, recent surgery, disabsortive syndrome, malignancies, under lipid-lowering therapy, unable or unwilling to participate, or with less than 80% adherence to phytosterols

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change in total and LDL-cholesterol | 12 weeks
  Phytosterol suplementation can reduce by 5-10% plasma levels of total- and LDL-cholesterol

SECONDARY OUTCOMES:
Change in LDL subfractions | 12 weeks
  Phytosterol suplementation can modify LDL subfractions
Change in HDL subfractions | 12 weeks
  Phytosterol suplementation can modify HDL subfractions
Improvement on quality of LDL particle | 12 weeks
  Phytosterol supplementation can improve the quality of LDL particle

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Izar, M.D., Ph.D., Principal Investigator — Federal University of São Paulo
Locations (2):
- Brazil (2):
  - University of Sao Paulo, São Paulo, Other
  - Federal University of Sao Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request.
Supporting Information: Study Protocol, SAP
Time Frame: After publication, and for one year.
Access Criteria: Upon request

REFERENCES:
- [Derived] Machado VA, Santisteban ARN, Martins CM, Damasceno NRT, Fonseca FA, Neto AMF, Izar MC. Effects of phytosterol supplementation on lipoprotein subfractions and LDL particle quality. Sci Rep. 2024 May 15;14(1):11108. doi: 10.1038/s41598-024-61897-4. PMID 38750162